CLINICAL TRIAL: NCT00396383
Title: Treatment With AMD3100 in Multiple Myeloma Patients to Mobilize Peripheral Blood Progenitor Cells For Collection and for Transplantation
Brief Title: Treatment With AMD3100 (Plerixafor) in MM Patients to Mobilize PBCs For Collection and for Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient cell mobilization for tandem transplants
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: AnorMED (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2108
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Stem cell mobilization; apheresis
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants with Multiple Myeloma (MM) (Experimental): Participants with MM who were eligible for autologous peripheral blood stem cell transplantation.
  Interventions: Drug: plerixafor

INTERVENTIONS:
Drug: plerixafor — Participants were given a 240 µg/kg dose of plerixafor by subcutaneous injection in the morning followed by apheresis 6 hours later. Daily treatment with plerixafor followed by apheresis was administered for up to 4 consecutive days or until 4*10^6 CD34+ cells/kg body weight had been collected.
  Other Names: Mozobil; AMD3100

SUMMARY:
This study will examine whether 240 µg/kg plerixafor given alone for up to 4 days is safe and well tolerated in multiple myeloma (MM) patients. In addition, this study determines if plerixafor alone can be used to mobilize peripheral blood progenitor cells (PBPCs) for transplantation in MM patients. The minimum number of CD34+ cells to collect is 2*10^6 CD34+ cells/kg and the target is ≧4*10^6 CD34+ cells/kg. Success of transplant engraftment will be measured by the number of days to polymorphonuclear leukocytes (PMN) and platelet (PLT) engraftment. Durability of transplant will be assessed for a minimum of one year.

DETAILED DESCRIPTION:
This study will examine whether 240 µg/kg plerixafor given alone for up to 4 days is safe and well tolerated in multiple myeloma (MM) patients. In addition, this study determines if 240 µg/kg plerixafor alone can be used to mobilize peripheral blood progenitor cells (PBPCs) for transplantation in MM patients. The minimum number of CD34+ cells to collect is 2*10^6 CD34+ cells/kg and the target is ≧4*10^6 CD34+ cells/kg. Success of transplant engraftment will be measured by the number of days to polymorphonuclear leukocytes (PMN) and platelet (PLT) engraftment. Durability of engraftment will be assessed for a minimum of one year.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM)
* Eligible for autologous transplantation
* Patients in first or second partial remission (PR) or complete remission (CR)
* Patients who have received ≦2000 rads of prior radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Recovered from all acute toxic effects of prior chemotherapy
* White blood cells (WBC) >3.0*10^9/l
* Absolute polymorphonuclear leucocyte (PMN) count >1.5*10^9/l
* Platelet (PLT) count > 150*10^9/l
* Serum creatinine ≦2.2 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 x upper limit of normal (ULN)
* Negative for HIV
* Signed informed consent
* Patients of childbearing potential agree to use an approved form of contraception

Exclusion Criteria:

* Patient received 2 or more alkylating agents, such as VBMCP (a combination of Vincristine, BCNU (Bis-Chloronitrosourea), Melphalan, Cyclophosphamide, and Prednisone)
* Patient received a total dose of ≧200 mg of prior melphalan
* A co-morbid condition which, in the view of the investigators, renders the patient at high risk from treatment complications
* Patient has failed previous collections or collection attempts
* A residual acute medical condition resulting from prior chemotherapy
* Brain metastases or carcinomatous meningitis
* Acute infection
* Fever (temperature >38 °C / 100.4 °F)
* Hypercalcemia (>1mg/dl above ULN)
* Positive pregnancy test in female patients
* Lactating females
* Patients of childbearing potential unwilling to implement adequate birth control
* Patients whose actual body weight exceeds 175% of their ideal body weight
* History of ventricular arrhythmias
* Patient received thalidomide within 10 days prior to receiving the first dose of plerixafor
* Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol or who are currently enrolled in another experimental protocol during the mobilization phase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Flomenberg N, Comenzo R, Badel K, Calandra G. Single agent AMD3100 mobilization of peripheral blood progenitor cells for autologous transplantation in patients with multiple myeloma (MM) [abstract]. Blood. Nov 16 2006;108(11 Pt 1):965a.
- [Result] Flomenberg N, Comenzo RL, Badel K, Calandra G. Plerixafor (Mozobil) alone to mobilize hematopoietic stem cells from multiple myeloma patients for autologous transplantation. Biol Blood Marrow Transplant. 2010 May;16(5):695-700. doi: 10.1016/j.bbmt.2009.12.538. Epub 2010 Jan 11. PMID 20067838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began in November 2004 and the study was terminated in May 2007. A total of 20 participants were planned for this study, however the study was terminated early because of insufficient mobilization of CD34+ cells after treatment with plerixafor alone for use in tandem transplants.
Groups:
- Participants With Multiple Myeloma (MM): Participants with MM who were eligible for autologous peripheral blood stem cell transplantation were given 240 µg/kg daily subcutaneous plerixafor for up to 4 days.
Period: Overall Study
Arm/Group | Participants With Multiple Myeloma (MM)
Started | 9
Completed | 6
Not Completed | 3
Not completed — Death | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved ≥4*10^6 CD34+ Cells/kg
Description: Number of participants achieving a target of ≥ 4*10^6 CD34+ cells/kg during apheresis for up to 4 consecutive days. Apheresis was performed six hours following treatment with plerixafor 240 µg/kg (alone). Target was calculated as the sum of all daily values collected from central laboratory data over up to 4 apheresis days.
Time Frame: Day 1 up to day 4
Population: All participants who received plerixafor
Measure: Number; unit: participants
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
participants
  Participants Who Achieved ≥4*10^6 cells | 4
  Participants Who Achieved <4*10^6 cells | 5

2. Primary Outcome: Participant Counts of Summarized Adverse Events (AE) During Treatment
Description: Participant counts of summarized adverse events (AEs) which occurred from the first dose of plerixafor up to the day prior to chemotherapy/ablative treatment. Events were graded according to World Health Organization criteria: Mild (awareness of sign or symptom, but easily tolerated), Moderate (discomfort enough to cause interference with usual activity), Severe (incapacitating with inability to work or do usual activity).
Time Frame: 1 month
Population: All participants who received plerixafor
Measure: Number; unit: participants
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
participants
  AE Severity (Mild) | 3
  AE Severity (Moderate) | 6
  AE Severity (Severe) | 0
  Life-threatening AE | 0
  AE Relationship to Drug (Not related) | 4
  AE Relationship to Drug (Probably not related) | 1
  AE Relationship to Drug (Possibly related) | 1
  AE Relationship to Drug (Probably related) | 3
  AE Relationship to Drug (Definitely related) | 0

3. Secondary Outcome: Number of Transplantations That Achieved Polymorphonuclear Leukocyte (PMN) Engraftment Grouped by Days to Engraftment
Description: Polymorphonuclear cell (PMN) engraftment was defined as a PMN count ≥ 0.5*10^9/L for 3 consecutive days or ≥ 1*10^9/L for 1 day. Days to engraftment corresponded to the first day that the criteria were met after transplantation.
Time Frame: Approximately 2 months
Population: Intent to treat population includes participants who received plerixafor and underwent transplantation. One participant had two transplants.
Measure: Number; unit: transplantations
Units Other Than Participants: transplantations
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
Number analyzed (transplantations) | 10
transplantations
  <= Day 12 post transplant | 10
  Day 13 to 21 post transplant | 0
  >= Day 22 post transplant | 0

4. Secondary Outcome: Number of Transplantations That Achieved Platelet (PLT) Engraftment Grouped by Days to Engraftment
Description: Platelet (PLT) engraftment was defined as a PLT count of ≥ 20*10^9/L for 7 days without transfusion. Days to engraftment corresponded to the first day that the criteria were met after transplantation.
Time Frame: Approximately 2 months
Population: Intent to treat population includes participants who received plerixafor and underwent transplantation. One participant had two transplants. One participant did not have PLT samples collected (included as 'unknown' in data table).
Measure: Number; unit: transplantations
Units Other Than Participants: transplantations
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
Number analyzed (transplantations) | 10
transplantations
  <= Day 12 post transplant | 0
  Day 13 to 21 post transplant | 6
  >= Day 22 post transplant | 3
  Unknown | 1

5. Secondary Outcome: Number of Participants With a Durable Graft at 12 Months Post Transplantation
Description: Graft durability was assessed by the Investigator based on complete blood count (CBC) and differential analyses at 12 months post transplantation.
Time Frame: Approximately month 13
Population: Intent to treat population includes participants who received plerixafor, underwent transplantation, and were evaluable 12 months post transplant.
Measure: Number; unit: participants
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 6
participants | 6

6. Post Hoc Outcome: Number of Participants Who Achieved ≥2*10^6 CD34+ Cells/kg
Description: Number of participants achieving ≥ 2*10^6 CD34+ cells/kg during apheresis for up to 4 consecutive days. Apheresis was performed six hours following treatment with plerixafor 240 µg/kg (alone). Total was calculated as the sum of all daily values collected from central laboratory data over up to 4 apheresis days.
Time Frame: Day 1 up to day 4
Population: All participants who received plerixafor
Measure: Number; unit: participants
Arm/Group | Participants With Multiple Myeloma (MM)
Number analyzed (Participants) | 9
participants | 9

ADVERSE EVENTS:
Time Frame: The first day of plerixafor administration up to the day prior to chemotherapy/ablative treatment.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Each AE table includes events, regardless of reported relationship to study treatment or grade.
Arm/Group | Participants With Multiple Myeloma (MM)
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Multiple Myeloma (MM) (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Catheter site erythema (General disorders) | 1
Catheter site related reaction (General disorders) | 1
Infusion site bruising (General disorders) | 1
Injection site erythema (General disorders) | 3
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Heart rate irregular (Investigations) | 1
Platelet count decreased (Investigations) | 1
Syphilis test positive (Investigations) | 1 — Female- history of syphilis- previous treatment unknown. On Day 3 plerixafor therapy, tested positive for (1:16) rapid plasma reagin titer. Doxycycline given for 5 weeks. No post-treatment titer and no comment made at her 12-month follow-up visit.
Hypokalaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study had limited enrollment prior to termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.